CLINICAL TRIAL: NCT03140735
Title: Interest of Pulse Wave Velocity Measurement as a Predictor of Severity of Aortic Stenosis
Acronym: VOPRABIO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2016_843_0035
Record Dates: First submitted 2017-04-14; First posted 2017-05-04 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Pulse Wave; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group of 150 heart disease-free individuals (Other)
  Interventions: Other: Control group without heart disease
- Patients with aortic sclerosis (Other)
  Interventions: Other: Study the relationship between the arterial rigidity of large vessels and the presence and severity of degenerative aortic constriction
- Patients with moderate aortic stenting (RA) (Other)
  Interventions: Other: Study the relationship between the arterial rigidity of large vessels and the presence and severity of degenerative aortic constriction
- Patients with Serious Aortic Retention (Other)
  Interventions: Other: Study the relationship between the arterial rigidity of large vessels and the presence and severity of degenerative aortic constriction

INTERVENTIONS:
Other: Study the relationship between the arterial rigidity of large vessels and the presence and severity of degenerative aortic constriction — Study the relationship between the arterial rigidity of large vessels and the presence and severity of degenerative aortic constriction
  Arms: Patients with Serious Aortic Retention; Patients with aortic sclerosis; Patients with moderate aortic stenting (RA)
Other: Control group without heart disease — Control group without heart disease
  Arms: Control group of 150 heart disease-free individuals

SUMMARY:
Aortic valve pathology is the third most common cardiovascular disease after coronary artery disease and hypertension, which is responsible for severe morbidity and mortality in elderly patients and requires surgical treatment in its most severe form of progression. The purpose of this study is to find a link between arterial stiffness and degenerative aortic stenosis. If this link is established, arterial stiffness may become a medical therapeutic target in order to delay the evolution of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, without legal protection (guardianship or curatorship),
* Stable hemodynamic status.
* Affiliation to a social security scheme

Exclusion Criteria:

* Hemodynamically unstable patients: Systolic PA <10 cmHg, rapid peripheral pulse and spinning, mottling, obnubilation, oliguria, sweating, coma
* History of significant valvulopathy other than an aortic stenosis,
* Pregnancy.
* Patient under tutelage or curatelle or deprived of public right.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Analysis of echocardiographic measurements of possible differences between average VOP and Sao i in terms of RA severities | 10 years
  Analysis of echocardiographic measurements of possible differences between average VOP and Sao i in terms of RA severities

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France